CLINICAL TRIAL: NCT03543813
Title: A Phase 1-2, First-in-Human Study of CX-2029 in Adults With Metastatic or Locally Advanced Unresectable Solid Tumors or Diffuse Large B-cell Lymphomas (PROCLAIM-CX-2029)
Brief Title: PROCLAIM-CX-2029: A Trial to Find Safe and Active Doses of an Investigational Drug CX-2029 for Patients With Solid Tumors or DLBCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CytomX Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMX-M-2029-001
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor, Adult; Head and Neck Cancer; Non Small Cell Lung Cancer; Diffuse Large B Cell Lymphoma; Esophageal Cancer
Keywords: cancer; solid tumor; DLBCL; CX-2029; PROBODY™ Therapeutic; Drug Conjugate; Antibody drug conjugate; CD71; Transferrin receptor 1
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Lymphoma, Large B-Cell, Diffuse; Esophageal Neoplasms; Neoplasms | interventions — CX-2029

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CX-2029 Escalation (Experimental): Dose Escalation and Determination
  Interventions: Drug: CX-2029
- CX-2029 Biomarker (Experimental): Characterization of CX-2029 in the tumor microenvironment in subjects with select tumor types
  Interventions: Drug: CX-2029
- CX-2029 Expansion (Experimental): Evaluate antitumor activity of CX-2029
  Interventions: Drug: CX-2029

INTERVENTIONS:
Drug: CX-2029 — CX-2029 Monotherapy

SUMMARY:
The purpose of this first-in-human study of CX-2029 is to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and antitumor activity of CX-2029 in adult subjects with metastatic or locally advanced unresectable solid tumors or diffuse large B-cell lymphoma (DLBCL). The antitumor activity of CX-2029 will be evaluated in subjects with head and neck squamous cell carcinoma (HNSCC), DLBCL, non-small cell lung cancer (NSCLC) (squamous cell histology only), or esophageal (esophageal adenocarcinoma [EAC], esophageal squamous cell carcinoma [ESCC], or gastroesophageal [GE] junction) cancer.

PROCLAIM: PRObody CLinical Assessment In Man CX-2029 clinical trial 001

PROBODY is a trademark of CytomX Therapeutics, Inc

DETAILED DESCRIPTION:
This is an open-label, Phase 1-2, first-in-human study for CX-2029 in subjects with metastatic or locally advanced unresectable solid tumors or Diffuse large B-cell lymphoma (DLBCL) without approved life-prolonging treatment options for their malignancy.

The study is divided into 3 parts (arms), as follows:

* Part A: Dose escalation and determination of the Maximum tolerated dose (MTD) and/or Recommended Phase 2 dose (RP2D)
* Part B: Characterization of CX-2029 in the Tumor microenvironment (TME) in subjects with select tumor types using previously cleared dose levels from Part A
* Part C: Expansions in select tumor types at the MTD/RP2D as established in Part A

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of metastatic or locally advanced unresectable tumors
2. Patients demonstrating disease progression after treatment with approved therapies that are known to confer life-prolonging benefit, or who are intolerant to or have declined treatment
3. Agreement to provide mandatory archival tissue or fresh biopsy
4. At least 18 years of age
5. For Arm A, histologically or cytologically confirmed metastatic or locally advanced unresectable solid tumor
6. For Arms B and C, histologically or cytologically confirmed metastatic or locally advanced unresectable HNSCC, DLBCL, NSCLC (squamous cell histology only), or esophageal (EAC, ESCC, or GE junction) cancer
7. Additional inclusion criteria may apply

Exclusion Criteria:

1. Neuropathy > Grade 1
2. Serious concurrent illness, including clinically relevant active infection
3. Clinically significant iron metabolism disorders (eg, sickle cell anemia)
4. Significant cardiac disease such as recent myocardial infarction
5. History of multiple sclerosis or other demyelinating disease, Eaton-Lambert syndrome (para-neoplastic syndrome), history of hemorrhagic or ischemic stroke within the last 6 months, or alcoholic liver disease;
6. Non-healing wound(s) or ulcer(s) except for ulcerative lesions caused by the underlying neoplasm;
7. History of severe allergic or anaphylactic reactions to previous monoclonal antibody therapy;
8. Currently receiving anticoagulation therapy with warfarin;
9. Major surgery (requiring general anesthesia) within 3 months prior to dosing.
10. Hepatic impairment which is moderate (Child-Pugh B) or severe (Child-Pugh C)
11. Transfusion dependent anemia with transfusion dependency of ≥3 months
12. Use of iron chelators
13. Additional exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The number of subjects experiencing a dose-limiting toxicity at various dose levels when given CX-2029 as a monotherapy | 21 days (dose-limiting toxicity period)

SECONDARY OUTCOMES:
The percentage of subjects experiencing anti-cancer activity (ORR) at various dose levels when given CX-2029 as a monotherapy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Monika Vainorius, M.D., Study Director — CytomX Therapeutics, Inc.
Locations (25):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - University of Southern California, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists, Lake Mary, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Forrest General Cancer Center, Hattiesburg, Mississippi
  - Washington University - St. Louis, St Louis, Missouri
  - New York University (NYU) Clinical Cancer Center, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- South Korea (3):
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Kangbuk Samsung Hospital, Seoul, Jongno-gu
  - Severance Hospital- Yonsei Cancer Center, Seoul, Seodaemun-gu
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario La Paz, Servicio de Oncología, Madrid
  - Centro Integral Oncologico Clara Campal, START Madrid, Madrid
  - Hospital Universitario Quiron de Madrid, Madrid
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Withington, Manchester Greater
  - Beatson, West of Scotland Cancer Centre, Glasgow

IPD SHARING:
Plan to Share IPD: No